CLINICAL TRIAL: NCT06674083
Title: Reliability of the Gyko Inertial Sensor System in Evaluating Jumping and Postural Stability Parameters in Healthy Adults
Status: Not yet recruiting | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Birgül Dıngırdan, Research Assisstant, Hacettepe University
Other Study IDs: Sakarya University of Applied; E-26428519-050.99-145546 (Other: Sakarya University of Applied Sciences)
Record Dates: First submitted 2024-11-03; First posted 2024-11-05 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Assessment, Self; Sports Physical Therapy
Keywords: Gyko inertial sensor system; Jump; Reliability; Postural stability

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy adults: Inclusion criteria for participants are as follows: being between the ages of 18 and 30, having no balance issues (such as vertigo) that could affect assessments, and having no health problems that would interfere with understanding the assessments.

SUMMARY:
The aim of the study is to examine the Gyko inertial sensor system in healthy adults. In the study, jump and postural control parameters are assessed with a one-week interval. To evaluate intra-rater reliability, ICC, SEM, and MDC values will be calculated.

DETAILED DESCRIPTION:
The Gyko inertial sensor system is a lightweight and portable device that applies protocols for assessing and monitoring joint function, muscle strength, jump, and postural stability parameters during the rehabilitation of a specific musculoskeletal region. Previous studies have evaluated the validity of Gyko in assessing vertical jump height in female sub-elite soccer players and its reliability in evaluating postural stability in healthy, non-athletic adults. However, the findings regarding both the validity and reliability of the device have been limited.

Our aim in this study is to evaluate the reliability of the Gyko inertial sensor system, an affordable and accessible tool that facilitates the assessment and monitoring of jump and postural stability parameters in healthy adults. If the study confirms the reliability of the Gyko device in evaluating these parameters, it could be used by clinicians, therapists, researchers, and/or coaches as a targeted alternative to gold standard methods for assessing jump and postural stability parameters in healthy adults.

Hypotheses:

H0: The use of the Gyko inertial sensor system is not reliable for assessing jump and postural control parameters in healthy adults.

H1: The use of the Gyko inertial sensor system is reliable for assessing jump performance in healthy adults.

H2: The use of the Gyko inertial sensor system is reliable for assessing postural control in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* being between the ages of 18 and 35
* having no balance issues (such as vertigo) that could affect assessments
* having no health problems that would interfere with understanding the assessments.

Exclusion Criteria:

* Having known neurological, rheumatological, or musculoskeletal system problems.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Sample size calculations were based on the ICC (0.81-0.87) data for jump parameters obtained from the reference study. Accordingly, the minimum acceptable reliability (ICC) (ρ0) was set at 0.70, with the expected reliability (ICC) (ρ1) at 0.85, considering 80% power and a significance level of 0.05. As a result of the power analysis, it was determined that at least 50 participants should be included in the study. Considering a 10% possibility of separation in test-retest for the participants, it was decided to include 55 individuals.
Sampling Method: Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
The reliability of the jump and postural stability reliability with Gyko inertial system | two weeks
  Assessments will be repeated one week apart to evaluate the reliability of the Gyko inertial system in postural stability and jump performance parameters. Jump and postural stability assessment with Gyko inertial system.